CLINICAL TRIAL: NCT03605134
Title: The Impact of Routine Measurement of Cardiac Troponin (hsTnT) on Outcome in Elderly Patients Undergoing Major Surgery
Status: Terminated | Type: Observational
Why Stopped: Not enough patient recruited
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: Troponin
Record Dates: First submitted 2018-06-28; First posted 2018-07-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Surgery--Complications; Mortality; Elderly
Keywords: troponin; diastolic function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample: High sensitive Troponin T
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: level of cardiac troponin and diastolic function assessment by means of transthoracic echocardiography
  Interventions: Diagnostic Test: level of cardiac troponin; Diagnostic Test: diastolic function assessment

INTERVENTIONS:
Diagnostic Test: level of cardiac troponin — blood test
Diagnostic Test: diastolic function assessment — transthoracic echocardiography

SUMMARY:
To document levels of cardiac troponin hsTnT in patients above 75y undergoing high risk surgery and the relationship between elevated levels and outcome in terms of hospital stay and 30 day mortality.

DETAILED DESCRIPTION:
Elevated troponin (Tn) hsTnT levels occur as a result of myocardial damage and are used in the diagnosis of myocardial infarction (MI). However, there are multiple different causes that also result in abnormal Tn levels, such as direct myocardial-cell injury, impaired renal excretion and sepsis. Because of this, elevated Tn level is a common finding in hospitalized patients.

Several studies on patients admitted to the intensive care unit (ICU) without MI show that Tn elevation is a mortality risk factor and an independent predictor of hospital mortality.

Up till now it is not yet known if the routine measurement of Tn in elderly patients undergoing surgery can significantly improve their outcome and that is the primary aim of this study. In addition, it is not known what the impact could be if a diastolic function assessment could be performed peri-operatively.

This study will examine the correlation between elevated Tn levels in elderly patients undergoing major surgery and their short-term outcome (in-hospital). Before and immediately after surgery, diastolic function will be assessed by means of transthoracic echocardiography (TTE).

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥75 y undergoing elective and major surgery till we have collected an entire dataset of 100 patients.
* Only those patients will be included who are planned for elective and major surgery.

Exclusion Criteria:

* Patients under the age of 75
* Intraoperative mortality
* Eye surgery
* Cardiac or thoracic surgery
* Patients undergoing surgery which is not withheld as major surgery
* For patients undergoing multiple surgeries for the same indication and during the same hospitalization, only the first surgery will be included

Ages: 75 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All surgical patients above 75 years old
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-08-07 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
surgical mortality | 30 days
  30 days mortality

SECONDARY OUTCOMES:
diastolic function | 3 days
  transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: jan Poelaert, PhD, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Patrice Forget, PhD, MD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium